CLINICAL TRIAL: NCT05986110
Title: Analysis of the Results Obtained in the Regular Clinical Practice of a Clinical Ultrasound Classroom For Primary Care Physicians As a Formative Intervention System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacion para la Investigacion y Formacion en Ciencias de la Salud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IBYAP22/00008
Record Dates: First submitted 2023-06-29; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-06

CONDITIONS: Family Medicine; Clinical Ultrasound; Primary Care
Keywords: Family medicine; Clinical ultrasound; Primary care; Resolution improvement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Procedure: A training intervention on clinical ultrasound
- Control Group (No Intervention)

INTERVENTIONS:
Procedure: A training intervention on clinical ultrasound — To train 20 primary care family doctors in clinical ultrasound so that they have greater power of resolution and allow them to limit the diagnostic and surgical times on the waiting lists of their patients.
  Arms: Intervention Group

SUMMARY:
The objectives of the project are to evaluate the theoretical-practical knowledge acquired and the degree of satisfaction of a methodology based on theoretical-practical training in abdominal and thyroid clinical ultrasound of family doctors, in the urban area of Primary Health Care, and to evaluate the benefit obtained by patients over 60 years of age included in the program, analyzing the degree of satisfaction, resolution time of the reason for consultation and decrease in the number of referrals to the second level of care, analyzing the differences by gender.

DETAILED DESCRIPTION:
The objectives of the project are to evaluate the theoretical-practical knowledge acquired and the degree of satisfaction of a methodology based on theoretical-practical training in abdominal and thyroid clinical ultrasound of family doctors, in the urban area of Primary Health Care, and to evaluate the benefit obtained by patients over 60 years of age included in the program, analyzing the degree of satisfaction, resolution time of the reason for consultation and decrease in the number of referrals to the second level of care, analyzing the differences by gender.

The expected impact is that the doctors participating in the project learn to perform abdominal and thyroid ultrasound and continue to perform them during the year that their participation in the project lasts, and independently thereafter. In addition, this will allow the reduction of interconsultations to the specialized care and emergencies of their patients whose primary care physicians perform ultrasound scans in their health center.

Its application in clinical practice will be reflected because doctors who perform ultrasound scans in their primary care centers will increase their diagnostic certainty in real consultation time on many occasions, thereby reducing interconsultations at the second level of care, and when they have to refer a patient at this level, they will do so in a more documented manner.

ELIGIBILITY:
Inclusion Criteria:

* To work in selected health centers.
* To have assigned to more than 800 patients.
* Not have previous training in regulated clinical ultrasound.
* Sign a commitment to Attendance at least 80% of the training program sessions.
* Sign the informed consent.

Exclusion Criteria:

* Not meeting any of the inclusion criteria.
* Not signing the informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of knowledge and skills | 1 year
  An initial evaluation of knowledge will be carried out prior to the start of the training intervention, which will consist of 10 multiple choice questions with four possible answers with only 1 correct one (5 theoretical questions on the fundamentals and use of ultrasound, and interpretation of 5 images of pathologies or ultrasound anatomy). For the final evaluation, a new test will be carried out, with 10 questions similar to those of the initial test (5 theoretical questions and 5 common images).

CONTACTS AND LOCATIONS:
Locations (1):
- Primary Care Research Unit of Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No